CLINICAL TRIAL: NCT02222974
Title: A Single-blind, Placebo-controlled Single Increasing Dose Tolerance Study in Healthy Male Volunteers After Intravenous Administration of BIIR 561 CL (Dosage: 1mg/h - 175 mg/h), Infusion Time 1 Hour
Brief Title: Single Increasing Dose Tolerance Study in Healthy Male Volunteers of BIIR 561 CL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 600.1
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — irampanel

ARMS (2):
- BIIR 561 CL (Experimental)
  Interventions: Drug: BIIR 561 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIR 561 CL
  Arms: BIIR 561 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to obtain information about safety, tolerability and pharmacokinetics of BIIR 561 CL after single intravenous administration of increasing doses in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age 21 to 50 years
* Broca index from -20% to +20%
* Written informed consent prior to admission to the study

Exclusion Criteria:

* Medical examination, laboratory tests or ECG judged by the investigator to differ significantly from normal clinical values
* Known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Known diseases of the central nervous system (CNS) (such as epilepsy), CNS trauma in their medical history or with psychiatric or neurological disorders
* Known history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Intake of any other drug which might influence the results of the trial during the week previous to the start of the study
* Participation in another study with an investigational drug within the last two - months preceding this study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Alcohol use of more than 60 g per day
* Drug dependency
* Excessive physical activities (e.g. competitive sports) within the last week before the study
* Blood donation within the last 4 weeks (>= 100 ml)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 1999-01; Primary Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 9 days after drug administration
Number of subjects with clinically significant findings in vital functions | up to 9 days after drug administration
  blood pressure, pulse rate, respiratory rate, oral body temperature
Number of subjects with clinically significant findings in ECG | up to 9 days after drug administration
Number of subjects with clinically significant findings in EEG | up to 24 hours after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 9 days after drug administration

SECONDARY OUTCOMES:
Area under the concentration time curve (AUC) | up to 24 hours after drug administration
Maximum drug plasma concentration (Cmax) | up to 24 hours after drug administration
Time to peak drug plasma concentration (tmax) | up to 24 hours after drug administration
Total mean residence time (MRTtot) | up to 24 hours after drug administration
Mean residence time of disposition (MRTdisp) | up to 24 hours after drug administration
Apparent terminal half-life (t1/2) | up to 24 hours after drug administration
Total clearance (CLtot) | up to 24 hours after drug administration
Volume of distribution during the terminal phase (Vz) | up to 24 hours after drug administration
Volume of distribution at steady state (Vss) | up to 24 hours after drug administration
Renal clearance (CLR) | up to 24 hours after drug administration
Amount excreted into urine (Ae) | up to 24 hours after drug administration